CLINICAL TRIAL: NCT04974996
Title: A Phase 1b, Open-Label, Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Antitumor Activity of Loncastuximab Tesirine in Combination With R-CHOP in Patients With Previously Untreated Diffuse Large B-cell Lymphoma (LOTIS-8)
Brief Title: A Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Antitumor Activity of Loncastuximab Tesirine in Combination With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Participants With Previously Untreated Diffuse Large B-cell Lymphoma (LOTIS-8)
Acronym: LOTIS-8
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to not proceed with study.
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-106
Record Dates: First submitted 2021-07-22; First posted 2021-07-23 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Untreated Diffuse Large B-Cell Lymphoma; DLBCL; Loncastuximab Tesirine
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — loncastuximab tesirine; Prednisone; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive escalating doses of loncastuximab tesirine (initial dose of 60 μg/kg and highest dose possibly tested of 150 µg/kg) in combination with R-CHOP (rituximab 375 mg/m^2, cyclophosphamide 750 mg/m^2, doxorubicin 50 mg/m^2, vincristine 1.4 mg/m^2, and prednisone 100 mg/day) according to a standard 3+3 dose escalation design. The dose escalation part will be completed once the maximum tolerated dose (MTD)/recommended dose for expansion (RDE) has been identified.
  Interventions: Drug: Loncastuximab tesirine; Drug: Prednisone; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine
- Part 2: Dose Expansion (Experimental): Participants will receive the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) of loncastuximab tesirine in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) as determined in Part 1.
  Interventions: Drug: Loncastuximab tesirine; Drug: Prednisone; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine

INTERVENTIONS:
Drug: Loncastuximab tesirine — Intravenous (IV) infusion
  Other Names: ADCT-402; ZYNLONTA
Drug: Prednisone — Orally via tablet or capsule
Drug: Rituximab — Intravenous (IV) infusion
Drug: Cyclophosphamide — Intravenous (IV) infusion
Drug: Doxorubicin — Intravenous (IV) infusion
Drug: Vincristine — Intravenous (IV) infusion

SUMMARY:
The primary objective of this study is to characterize the safety and tolerability of loncastuximab tesirine in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) chemotherapy, and identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) for the combination therapy.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multi-center study in participants with previously untreated DLBCL, with a dose escalation part followed by dose expansion part.

Participants will be treated by loncastuximab tesirine in combination with R CHOP.

The duration of the study participation for each participant is defined as the time from the date of signed written informed consent to the completion of the follow-up period, withdrawal of consent, lost to follow-up, or death, whichever occurs first.

The study will include a Screening Period (of up to 28 days), a Treatment Period of 6 cycles (cycles of 3 weeks), and a Follow-up Period (approximately every 12 week visits) for up to approximately 3 years from end-of-treatment (EOT).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any study procedures
2. Male or female participant aged 18 years or older
3. Pathologic diagnosis of diffuse large B-cell lymphoma (DLBCL), as defined by the 2016 World Health Organization classification (including participants with DLBCL transformed from indolent lymphoma), or high-grade B cell lymphoma
4. Measurable disease as defined by the 2014 Lugano Classification
5. Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue sample. (If tissue block is not available, slides from a FFPE block may be acceptable for eligibility upon consultation with the Sponsor)
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
7. Adequate organ function as defined by screening laboratory values within the following parameters:

   1. Absolute neutrophil count ≥1.5 × 10^3/μL (off growth factors at least 72 hours)
   2. Platelet count ≥75 × 10^3/μL without transfusion in the past 7 days
   3. Hemoglobin ≥9 g/dL (4.96 mmol/L), transfusion allowed
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and gamma glutamyl transferase (GGT) ≤2.5 × the upper limit of normal (ULN)
   5. Total bilirubin ≤1.5 × ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 × ULN)
   6. Calculated creatinine clearance >30 mL/min by the Cockcroft and Gault equation

   Note: A laboratory assessment may be repeated a maximum of two times during the Screening period to confirm eligibility.
8. Left ventricular ejection fraction (LVEF) of ≥50%, assessed by echocardiography or cardiac multi-gated acquisition (MUGA) scan
9. Women of childbearing potential (WOCBP) must agree to use a highly effective method of contraception from the time of giving informed consent until at least 9 months after the last dose of study drug. Men with female partners who are of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 6 months after the last dose of study drug.

Women of childbearing potential are defined as sexually mature women who have not undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or who have not been postmenopausal (i.e., who have not menstruated at all) for at least one year. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Highly effective forms of birth control are methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Highly effective forms of birth control include: hormonal contraceptives (oral, injectable, patch, intrauterine devices), male partner sterilization, or total abstinence from heterosexual intercourse, when this is the preferred and usual lifestyle of the participant.

Note: The double-barrier method (e.g., synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), periodic abstinence (such as calendar, symptothermal, post ovulation), withdrawal (coitus interruptus), lactational amenorrhea method, and spermicide-only are not acceptable as highly effective methods of contraception.

Exclusion Criteria:

1. Known history of hypersensitivity to or positive serum human anti-drug antibody (ADA) to a cluster of differentiation 19 (CD19) antibody
2. Previous therapy with loncastuximab tesirine, rituximab, anthracycline, or cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP)
3. Known history of hypersensitivity to any component of study treatment (loncastuximab tesirine and rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone [R-CHOP])
4. Previous treatment for aggressive lymphoma (with exception of short corticosteroid course [up to 7 days] for symptom management)
5. Contraindication to receive granulocyte colony stimulating factors
6. Human immunodeficiency virus (HIV) seropositive with any of the following:

   1. Cluster of differentiation 4 (CD4) + T-cell (CD4+) counts <350 cells/μL
   2. Acquired immunodeficiency syndrome-defining opportunistic infection within 12 months prior to screening
   3. Not on anti-retroviral therapy, or on anti-retroviral therapy for <4 weeks at the time of Screening
   4. HIV viral load ≥400 copies/mL
7. Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load
8. Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load
9. History of Stevens-Johnson syndrome or toxic epidermal necrolysis
10. Lymphoma with active central nervous system involvement at the time of Screening, including leptomeningeal disease
11. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
12. Breastfeeding or pregnant
13. Significant medical comorbidities, including but not limited to, uncontrolled hypertension (blood pressure [BP] ≥160/100 mmHg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to Screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes, or severe chronic pulmonary disease.
14. Active systemic bacterial, viral, fungal, or other infection requiring systemic treatment at the time of Screening
15. Major surgery, radiotherapy, chemotherapy, or other anti-neoplastic therapy within 14 days prior to start of study drug (Cycle 1 Day 1 [C1D1]; cycle is 21 days), except shorter if approved by the Sponsor
16. Use of any other experimental medication within 14 days prior to start of study drug (C1D1; cycle is 21 days)
17. Received live vaccine within 4 weeks of C1D1; cycle is 21 days
18. Congenital long measure between Q wave and T wave in the electrocardiogram (QT) syndrome or a corrected Fridericia correction of the QT measure (QTcF) interval of >480 ms at Screening (unless secondary to pacemaker or bundle branch block)
19. Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary
20. Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the participant inappropriate for study participation or put the participant at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-03-11 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience Dose Limiting Toxicities (DLTs) in Part 1 | Day 1 to Day 21 of Cycle 1, where a cycle is 21 days
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 up to End of Treatment (up to 30 days after last dose of study treatment in this study or start of a new anticancer therapy, whichever is earlier; approximately 20 weeks)
  Frequency and severity of TEAEs and treatment-emergent serious adverse events (SAEs), graded according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Delay | Day 1 up to approximately 18 weeks
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Interruption | Day 1 up to approximately 18 weeks
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Reduction | Day 1 up to approximately 18 weeks
Number of Participants Who Experience a Clinically Significant Change from Baseline in Safety Laboratory Values | Baseline (Day 1) to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Number of Participants Who Experience a Clinically Significant Change from Baseline in Vital Signs | Baseline (Day 1) to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Number of Participants Who Experience a Clinically Significant Change from Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline (Day 1) to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
  ECOG performance status will be measured on a scale from grades 0-5, where a higher grade indicates a worse outcome.
Number of Participants Who Experience a Clinically Significant Change from Baseline in 12-Lead Electrocardiograms (ECGs) | Baseline (Day 1) to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Number of Participants Who Experience a Clinically Significant Change from Baseline in Left Ventricular Ejection Fraction (LVEF) Assessments | Baseline (Screening) to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 3.5 years
Duration of Response (DOR) | Up to approximately 3.5 years
Progression Free Survival (PFS) | Up to approximately 3.5 years
Overall Survival (OS) | Up to approximately 3.5 years
Complete Response Rate | Up to approximately 3.5 years
Average Concentration of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Maximum Concentration (Cmax) of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Time to Maximum Concentration (Tmax) of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Area Under the Concentration-Time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Area Under the Concentration-Time Curve from Time Zero to the End of the Dosing Interval (AUCtau) of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Area Under the Concentration-Time Curve from Time Zero to Infinity (AUCinf) of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Apparent Terminal Elimination Half-Life (Thalf) of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Clearance of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Steady-State Volume of Distribution (Vss) of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Accumulation Index of Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)
Number of Participants With Anti-Drug Antibody (ADA) Titers to Loncastuximab Tesirine | Day 2 to End of Treatment (up to 30 days after last dose of study treatment; approximately 20 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No